CLINICAL TRIAL: NCT04831892
Title: The Effect of Isosorbide Diesters Based Moisturizer on Skin Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Sytheon Ltd. (Industry)
Responsible Party: Principal Investigator, Raja Sivamani, MD MS AP, Principal Investigator, Integrative Skin Science and Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: I20-ISO1
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Atopic Dermatitis
Keywords: eczema; skin; dermatology; isosorbide diesters; skin microbiome
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Moisturizer Containing Isosorbide Diesters and Colloidal Oatmeal (Experimental): Topical lotion containing isosorbide diesters and colloidal oatmeal to be applied to the entire body once daily.
  Interventions: Other: Moisturizer Containing Isosorbide Diesters and Colloidal Oatmeal
- Moisturizer containing colloidal oatmeal (Active Comparator): Topical moisturizer with colloidal oatmeal to be applied to the entire body once daily
  Interventions: Other: Moisturizer containing Colloidal Oatmeal only

INTERVENTIONS:
Other: Moisturizer Containing Isosorbide Diesters and Colloidal Oatmeal — Study lotion containing 0.1% colloidal oatmeal along with 4% HydraSynol® DOI (Isosorbide Dicaprylate) and 4% HydraSynol® IDL/(Isosorbide Disunflowerseedate)
  Arms: Moisturizer Containing Isosorbide Diesters and Colloidal Oatmeal
Other: Moisturizer containing Colloidal Oatmeal only — Vehicle lotion containing 0.1% colloidal oatmeal.
  Arms: Moisturizer containing colloidal oatmeal

SUMMARY:
The overall objective of this study is to assess how a natural ingredient, isosorbide diesters (IDEAS), works in association with colloidal oatmeal for eczema.

DETAILED DESCRIPTION:
The topical therapy of eczema largely focuses on the use of topical medications but there is demand for topical moisturizers and ingredients that can reduce the need for topical steroids. The goal of this study is to assess the use of a natural ingredient, isosorbide diesters (IDEAS), for eczema and if it can reduce the need for the use of topical steroids.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or over
* Subjects with a diagnosis of mild to moderate eczema with a SCORAD between 1-50.

Exclusion Criteria:

* Individuals who have a known allergy to isosorbide diesters.
* Individuals who have solely hand and/or foot eczema without evidence of eczema anywhere else on their body.
* Individuals who have been on topical calcineurin inhibitors or crisaborole to the predetermined areas within two weeks of initiation of participation or unwilling to undergo a washout period.
* Subjects with an ongoing secondary infection of the skin.
* Subjects who are on systemic therapy or who need systemic therapy at the discretion of the investigator. Systemic therapies include cyclosporine, systemic steroids, methotrexate, and dupilumab. Subjects who have been on cyclosporine, systemic steroids, or methotrexate in the month prior to initiation of study intervention or are unwilling to undergo a washout period. Subjects who have been on dupilumab in two months prior to initiation of study intervention or are unwilling to undergo a washout period.
* Subjects with a diagnosis of Scabies.
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
EASI75 | Week 4
  75% improvement in Eczema severity is assessed using the Eczema Area and Severity Index
Change in IVAS | 4 weeks
  Itch severity is assessed using the Itch Visual Analog Scale.

SECONDARY OUTCOMES:
Change in EASI score | Week 1
  Eczema severity is assessed using the Eczema Area and Severity Index.
Change in EASI score | Week 5
  Eczema severity is assessed using the Eczema Area and Severity Index.
Change in IVAS | Week 1
  Itch severity is assessed using the Itch Visual Analog Scale.
Change in IVAS | Week 5
  Itch severity is assessed using the Itch Visual Analog Scale.
Change in TEWL | Week 1
  Transepidermal water loss (TEWL) is measured with a skin vapometer.
Change in TEWL | Week 4
  Transepidermal water loss (TEWL) is measured with a skin vapometer.
Change in TEWL | Week 5
  Transepidermal water loss (TEWL) is measured with a skin vapometer.
Change in skin hydration level | Week 1
  Skin hydration levels are measured using a moisture meter.
Change in skin hydration level | Week 4
  Skin hydration levels are measured using a moisture meter.
Change in skin hydration level | Week 5
  Skin hydration levels are measured using a moisture meter.
Change in DLQI survey responses | Week 1
  Self-reported quality of life through the Dermatology Life Quality Index, a survey completed by subjects.
Change in DLQI survey responses | Week 4
  Self-reported quality of life through the Dermatology Life Quality Index, a survey completed by subjects.
Change in DLQI survey responses | Week 5
  Self-reported quality of life through the Dermatology Life Quality Index, a survey completed by subjects.
Change in relative abundance of S. aureus | 4 weeks
  Skin microbiome related measurement of S. aureus relative abundance

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

REFERENCES:
- [Derived] Nadora D, Burney W, Chaudhuri RK, Galati A, Min M, Fong S, Lo K, Chambers CJ, Sivamani RK. Prospective Randomized Double-Blind Vehicle-Controlled Study of Topical Coconut and Sunflower Seed Oil-Derived Isosorbide Diesters on Atopic Dermatitis. Dermatitis. 2024 Jan-Feb;35(S1):S62-S69. doi: 10.1089/derm.2023.0329. PMID 38394048